CLINICAL TRIAL: NCT07397169
Title: Adjustable Sockets for Veterans With Lower Limb Amputation: Patient Reported Outcomes and Within-socket Pressures
Brief Title: Adjustable Prosthetic Sockets
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRD2-010-25M; 1I01RD002103-01 (Other Grant/Funding Number: US Department of Veterans Affairs); 1924445 (Other: gov.irbnet.org)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Lower Extremity Amputation
Keywords: lower limb amputation; transtibial amputation; below knee amputation; prosthetic socket; prosthesis

STUDY DESIGN:
Intervention Model Description: Each participant will wear an instrumented adjustable prosthetic socket.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Adjustable prosthetic socket (Experimental): Participants will wear an adjustable prosthetic socket.
  Interventions: Device: Adjustable prosthetic socket

INTERVENTIONS:
Device: Adjustable prosthetic socket — The investigators will fabricate and assemble an adjustable prosthetic socket for each participant whose shape is a duplicate of their existing, as-prescribed prosthetic socket. We will add three adjustable panels to the prosthetic socket which will be located over the medial and lateral proximal tibia region and the posterior gastrocnemius region. The position of the panels will be adjustable in and out using a cable mechanism.

SUMMARY:
Each year, around 1500 Veterans join the 623,000 Americans who live with a lower limb amputation. Many of these Veterans choose the arduous path of rehabilitation to remain ambulatory, a process that includes the prescription of a lower limb prosthesis. Much relies on the goodness of fit of their prosthesis. A good fit feels comfortable and enables a variety of ambulatory activities. A poor fit results in discomfort, often accompanied by chronic skin issues, and activities of daily living are curtailed.

Conventional prosthetic sockets are custom-built by a skilled prosthetist, carefully formed to fit the Veteran's residual limb, and good fits can usually be obtained. These sockets are rigid, fixed shape structures with the robustness of a bulldozer, built for sustained, heavy-duty action. Unfortunately, the shape of an individual's residual limb can change over time, such that a good fit eventually becomes poor. One estimate suggests a new below-knee socket is needed every three and a half years. The expense of replacing sockets that no longer fit is not insignificant. Medicare expenditures for replacement of existing below-knee sockets and associated components were estimated at $50M in 2017. Importantly, Medicare is estimated to be only 20% of the market, suggesting the estimated expenditure for the entire population with lower limb amputations is likely to be meaningfully larger. A good fitting prosthesis that maintains its fit over time would serve Veterans well.

A potential solution that could make a good fit last longer is an adjustable prosthetic socket. While little evidence is available to support prescription practice, the Centers for Medicare and Medicaid Services (CMS) recently authorized reimbursement for adjustable prosthetic sockets, suggesting a compelling need for such a product.

To investigate the potential for deleterious effects and how Veterans might use adjustable prosthetic sockets, the aim of this research is to determine the pressure applied to the residual limb by an adjustable prosthetic socket during activities of varying intensity and the activities that induce adjustments.

A laboratory-based human subject experiment will be conducted using a custom sensor placed inside the adjustable panel of a study-provided adjustable prosthetic socket. Participants will acclimate to the adjustable prosthetic socket for two weeks in the field, then return to the laboratory to perform seven activities. The pressure inside the prosthesis will be measured during these activities. Participants will also report how tight their socket feels after each activity.

DETAILED DESCRIPTION:
Prosthetic sockets enabling ambulatory mobility of Veterans with lower limb amputation are typically rigid, overly strong structural elements of fixed shape that act as the interface between the body and the environment. A Veteran's prosthetic socket is bespoke; it is meant to fit one person and one person only.

Changes in fit after the provision of a prosthesis are more common than not. Changes related to body mass, muscle atrophy, or personal fitness can happen over months while changes due to diet or diabetic complications can happen over hours. If the mismatch in shape between the residual limb and socket is small, the Veteran can manage the difference by donning or doffing residual limb socks. The approach is not ideal as some patients are more inclined to adopt the practice than others. If the mismatch in shape is large, a new prosthetic socket is usually required. Whether small or large, failure to manage changes can negatively affect their use of the prosthesis and the health of their residual limb.

Despite its limitations, the fixed-shaped prosthetic socket has been the standard-of-care for decades. However, a potentially significant event occurred in April 2024 when the Centers for Medicare and Medicaid Services (CMS) authorized reimbursement for adjustable prosthetic sockets. While the new authorization enables payment for its provision, there is little evidence to aid patients, providers, and payers in understanding the potential outcomes of prescribing an adjustable prosthetic socket.

The purpose of this research is to discover how Veterans use adjustable prosthetic sockets by measuring the pressure applied to the residual limb by an adjustable prosthetic socket during activities of varying intensity and identify what activities might induce an adjustment. The investigators will recruit ambulatory Veterans with unilateral transtibial amputations (n = 25) and fit them with an adjustable prosthetic socket.

Participants will wear an instrumented adjustable prosthetic socket after wearing a non-instrumented duplicate adjustable prosthetic socket for two weeks. Participants will be allowed to walk about for 5 to 10 minutes while the research prosthetist checks the fit and alignment of the study prosthesis. Pressure measurements will then be collected while sitting, standing, and walking. The standing and walking activities will be performed in random order, interspersed with 1-minute seated rests where the participant will release the adjustable panel pressure. The walking trials will be performed on a treadmill.

* Seated rest 5 min
* Random order with 1 min seated rest between each:

  * Stand 1 min
  * Walk self-selected speed 1 min
  * Walk up 10% slope at self-selected speed 1 min
  * Walk down 10% slope at self-selected speed 1 min
  * Walk 15% faster than self-selected speed 1 min
  * Walk self-selected speed 10 min Just prior to the beginning of each activity, the participant will told what the next activity is and prompted to adjust their socket accordingly. Participants will also be free to make adjustments during an activity. In this situation, the duration of the activity will be extended such that 1 minute of activity remains at the new adjustment setting. At the end of each activity, tightness will be assessed using a survey question. Specifically, after each activity, the investigators will ask each participant to rate the tightness of their adjustable prosthetic socket at the moment on a 0 to 10 scale.

In general, the investigators hypothesize that the pressure applied to the residual limb will depend on the activity, as will the tightness.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with lower limb amputation
* have a unilateral transtibial amputation
* wear a prosthesis for at least 4 hours a day by self-report
* at least one-year post-amputation
* have a modular prosthesis that includes a four-bolt socket attachment
* can walk on a treadmill

Exclusion Criteria:

* have an improper fit and suspension with their current prosthesis, and a good fit cannot be achieved with clinical resources
* have current skin irritation or injury to the residual limb, osteoarthritis, injury, or pain that interferes with walking ability

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Distal end pressure while seated (5 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments
  A pressure transducer will record the distal end residual limb pressure while the participant is seated for 5 minutes. The first four minutes of data will be truncated. The remaining first and last fifteen seconds of the fifth minute will also be truncated. The mean pressure will be calculated from the remaining 30 seconds of each trial.
Distal end pressure while standing (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments
  A pressure transducer will record the distal end residual limb pressure while the participant stands for 1 minute. The first and last fifteen seconds will be truncated. The mean pressure will be calculated from the remaining 30 seconds of each trial.
Distal end pressure while walking at self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the distal end residual limb pressure while the participant walks at self-selected speed for 1 minute. The first and last fifteen seconds will be truncated. The mean peak pressure from each step with the prosthesis will be calculated from the remaining 30 seconds of each trial.
Distal end pressure while walking up 10% slope at self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the distal end residual limb pressure while the participant walks up 10% slope at self-selected speed for 1 minute. The first and last fifteen seconds will be truncated. The mean peak pressure from each step with the prosthesis will be calculated from the remaining 30 seconds of each trial.
Distal end pressure while walking down 10% slope at self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the distal end residual limb pressure while the participant walks down 10% slope at self-selected speed for 1 minute. The first and last fifteen seconds will be truncated. The mean peak pressure from each step with the prosthesis will be calculated from the remaining 30 seconds of each trial.
Distal end pressure while walking 15% faster than self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the distal end residual limb pressure while the participant walks 15% faster than self-selected speed for 1 minute. The first and last fifteen seconds will be truncated. The mean peak pressure from each step with the prosthesis will be calculated from the remaining 30 seconds of each trial.
Distal end pressure while walking at self-selected speed (10 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the distal end residual limb pressure while the participant walks at self-selected speed for 10 minutes. The first nine minutes of data will be truncated. The remaining first and last fifteen seconds of the tenth minute will also be truncated. The mean peak pressure from each step with the prosthesis will be calculated from the remaining 30 seconds of each trial.
Adjustable posterior panel pressure while seated (5 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the adjustable posterior panel pressure while the participant is seated for 5 minutes. The first four minutes of data will be truncated. The remaining first and last fifteen seconds of the fifth minute will also be truncated. The mean pressure will be calculated from the remaining 30 seconds of each trial.
Adjustable posterior panel pressure while standing (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the adjustable posterior panel pressure while the participant stands for 1 minute. The first and last fifteen seconds will be truncated. The mean pressure will be calculated from the remaining 30 seconds of each trial.
Adjustable posterior panel pressure while walking at self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the adjustable posterior panel pressure while the participant walks at self-selected speed for 1 minute. The first and last fifteen seconds will be truncated. The mean peak pressure from each step with the prosthesis will be calculated from the remaining 30 seconds of each trial.
Adjustable posterior panel pressure while walking up 10% slope at self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the adjustable posterior panel pressure while the participant walks up 10% slope at self-selected speed for 1 minute. The first and last fifteen seconds will be truncated. The mean peak pressure from each step with the prosthesis will be calculated from the remaining 30 seconds of each trial.
Adjustable posterior panel pressure while walking down 10% slope at self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the adjustable posterior panel pressure while the participant walks down 10% slope at self-selected speed for 1 minute. The first and last fifteen seconds will be truncated. The mean peak pressure from each step with the prosthesis will be calculated from the remaining 30 seconds of each trial.
Adjustable posterior panel pressure while walking 15% faster than self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the adjustable posterior panel pressure while the participant walks 15% faster than self-selected speed for 1 minute. The first and last fifteen seconds will be truncated. The mean peak pressure from each step with the prosthesis will be calculated from the remaining 30 seconds of each trial.
Adjustable posterior panel pressure while walking at self-selected speed (10 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  A pressure transducer will record the adjustable posterior panel pressure while the participant walks at self-selected speed for 10 minutes. The first nine minutes of data will be truncated. The remaining first and last fifteen seconds of the tenth minute will also be truncated. The mean peak pressure from each step with the prosthesis will be calculated from the remaining 30 seconds of each trial.

SECONDARY OUTCOMES:
Tightness while seated (5 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  After each activity, the participant will rate the tightness of their adjustable prosthetic socket at the moment. On a 0 - 10 scale, if 0 represents the loosest socket fit that can be imagined, and 10 represents the tightest socket fit that can be imaged, what score represents the socket tightness at the moment?
Tightness while standing (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  After each activity, the participant will rate the tightness of their adjustable prosthetic socket at the moment. On a 0 - 10 scale, if 0 represents the loosest socket fit that can be imagined, and 10 represents the tightest socket fit that can be imaged, what score represents the socket tightness at the moment?
Tightness while walking at self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  After each activity, the participant will rate the tightness of their adjustable prosthetic socket at the moment. On a 0 - 10 scale, if 0 represents the loosest socket fit that can be imagined, and 10 represents the tightest socket fit that can be imaged, what score represents the socket tightness at the moment?
Tightness while walking up 10% slope at self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  After each activity, the participant will rate the tightness of their adjustable prosthetic socket at the moment. On a 0 - 10 scale, if 0 represents the loosest socket fit that can be imagined, and 10 represents the tightest socket fit that can be imaged, what score represents the socket tightness at the moment?
Tightness while walking down 10% slope at self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  After each activity, the participant will rate the tightness of their adjustable prosthetic socket at the moment. On a 0 - 10 scale, if 0 represents the loosest socket fit that can be imagined, and 10 represents the tightest socket fit that can be imaged, what score represents the socket tightness at the moment?
Tightness while walking 15% faster than self-selected speed (1 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  After each activity, the participant will rate the tightness of their adjustable prosthetic socket at the moment. On a 0 - 10 scale, if 0 represents the loosest socket fit that can be imagined, and 10 represents the tightest socket fit that can be imaged, what score represents the socket tightness at the moment?
Tightness while walking at self-selected speed (10 min bout) | After a two-week acclimation period where the participant wears an adjustable prosthetic socket in the home, community, and work environments.
  After each activity, the participant will rate the tightness of their adjustable prosthetic socket at the moment. On a 0 - 10 scale, if 0 represents the loosest socket fit that can be imagined, and 10 represents the tightest socket fit that can be imaged, what score represents the socket tightness at the moment?

CONTACTS AND LOCATIONS:
Overall Officials: Glenn K Klute, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the proposed research will be shared outside VA. A de-identified, anonymized dataset will be created and available to the public via a VA authorized website. Where possible, the investigators will work with manuscript publishers to link the final study data sets as an appendix to published manuscripts. By providing de-identified datasets in open file formats (e.g., .txt, .xls, .mat) along with clearly documented instructions for processing, interested recipients will be able to reproduce and build on the same techniques which the investigators will outline in our publications. A public release identifier for each subject's data (e.g., APS_001, APS_002) will be created and randomly paired with de-identified study data. Data will consist of subject demographics, test, and questionnaire results. There will be no tractable way to re-match these data to the subject. Our methods will be verified by the VAPSHCS Privacy Officer.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within six months of publication of final study findings.
Access Criteria: Open access through PubMed Central, SimTK, PhysioNet, or other similar open-source data repository websites. The study protocol, statistical analysis plan, and the informed consent form will be shared on clinicaltrials.gov.